CLINICAL TRIAL: NCT02008760
Title: Survey of Chronic Pain Patients' Self-rated Quality of Life, ADL Function and Pain Before and After Intervention With Omega 3 Fatty Acids From Krill With Vitamin D3
Brief Title: QOL, ADL and Pain Before and After Intervention With N3 From Krill With D3.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospitalet Valdemar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJ-327
Record Dates: First submitted 2013-12-07; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Quality of Life; Pain
Keywords: pain; quality of life; ADL; DOLO test; compliance; D3
MeSH Terms: conditions — Pain; Patient Compliance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vegetable oil with betacarotene (Placebo Comparator): 4 capsules vegetable oil with betacarotene
- krill and vitamin D3 (Active Comparator): krill and vitamin D3. (72 mg), four capsules daily
  Interventions: Dietary Supplement: Omega Krill with D3

INTERVENTIONS:
Dietary Supplement: Omega Krill with D3
  Arms: krill and vitamin D3

SUMMARY:
The aim of this project is investigation of patients' with chronic pain self-rated quality of life, ADL function and level of pain before and after 3 months of intervention with N-3 fatty acids from krill in combination with vitamin D3. Furthermore, the compliance of the patients and the effect of the intervention on the patients' vitamin D status and cardiovascular risk factors are studied.

ELIGIBILITY:
Inclusion Criteria:

* 18 year +
* can read and understand danish

Exclusion Criteria:

* shellfish allergy
* intake of anticoagulants and vitamin D
* pacemaker
* participating other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
ADL function on a scale 0-11 | february 2013-february 2014
pain on a scale 0-100 mm | february 2013-february 2014
Quality of life on a scale 0-100 | february 2013-february 2014

SECONDARY OUTCOMES:
compliance in % | february 2013-february 2014
changes at D3 levels | february 2013-february 2014

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Nielsen, C physician, Principal Investigator — Hospitalet Valdemar
Locations (1):
- Hospitalet Valdemar, Ringsted, Denmark